CLINICAL TRIAL: NCT02836379
Title: Quality of Life Study in Patients With Breakthrough Cancer Pain Treated in Radiation Oncology Services With Palliative Intent
Brief Title: Quality of Life Study Breakthrough Cancer Pain Treated in Radiation Oncology Services With Palliative Intent
Acronym: CAVIDIOR
Status: Completed | Type: Observational
Sponsor: Angelini Farmacéutica (Industry)
Responsible Party: Sponsor
Other Study IDs: ANG-DOL-2016-01 (CAVIDIOR)
Record Dates: First submitted 2016-07-11; First posted 2016-07-19 (Estimated); Last update posted 2018-03-05 (Actual); Status verified 2018-03

CONDITIONS: Breakthrough Pain
Keywords: Breakthrough Cancer Pain; Quality of life; Radiotherapy
MeSH Terms: conditions — Breakthrough Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Breakthrough Cancer Pain: No intervention (Non-interventional study)
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
In the context of radiotherapy, control of breakthrough pain represents a special challenge. Patients undergoing radiotherapy may experience different situations of pain that may be due to the need to remain immobilized during radiotherapy session, the need to wear an immobilization mask (head and neck cancer), the odynophagia caused by mucositis, defecation after the development of proctitis, or sudden pain during the night causing sleep disturbances.

In a survey conducted in radiation oncology services more than half of patients treated with radiotherapy experienced pain, and 39% of patients reported that their pain was not treated properly. This situation may increase the patient's anxiety, dissatisfaction with treatment, affect their quality of life and can even come to refuse radiotherapy treatment.

This post-authorization observational study will assess the quality of life of cancer patients with breakthrough cancer pain treated in radiotherapy services in Spanish hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years
* Cancer Patients
* Patients attended in radiation oncology consultations with palliative intent
* Life expectancy > 6 months
* Written informed consent
* Patients with baseline controlled cancer pain with opioids who are diagnosed of breakthrough cancer pain by Davies algorithm

Exclusion Criteria:

* Untreated patients with opioids for baseline pain
* Patients who are not opioid tolerant
* Serious psychiatric disorder or any disease or condition that prevents the collection of data
* Patients with evidence of opioid addiction or history of drug or alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with breakthrough cancer pain treated in Radiation Oncology services with palliative intent will be included
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2016-07-08 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Change in quality of life according SF-12 questionnaire | Baseline and 4-6 weeks (estimated end of radiotherapy treatment)
  Change in punctuation of the SF-12 questionnaire between end of radiotherapy treatment and baseline.

SECONDARY OUTCOMES:
Percentage of patients with neuropathic, visceral, somatic and mixed pain | Baseline (the day that patient sign the informed consent form)
  Percentage of patients with neuropathic, visceral, somatic and mixed pain
Comorbidities associated with patients | Baseline (the day that patient sign the informed consent form)
  Percentage of patients with each comorbidity
Mean time to relief of breakthrough pain | Up to 6 weeks, from date of inclusion until the end of radiotherapy treatment
  Time from the start of the episode until the relief of breakthrough pain
Mean duration of the episodes of breakthrough pain | Up to 6 weeks, from date of inclusion until the end of radiotherapy treatment
  Time from the start of the episode until the pain ends
Clinical Global improvement | 4-6 weeks (estimated end of radiotherapy treatment)
  Number of patients indicating each of the possible answers of the Clinical Global Impression of improvement scale
Patient Global improvement | 4-6 weeks (estimated end of radiotherapy treatment)
  Number of patients indicating each of the possible answers of the Patient Global Impression of improvement scale
Change in assessment (percentage) of family claudication | Baseline and 4-6 weeks (estimated end of radiotherapy treatment)
  Difference in percentage of patients with punctuation ≥ 17 points at end of radiotherapy treatment and baseline.
Change in mean Intensity of breakthrough cancer pain at each study visit | Up to 6 weeks, from date of inclusion until the end of radiotherapy treatment
  Intensity of breakthrough cancer pain assessed with a Visual Analog Scale (VAS). VAS will be compared at each study visit.
Change in MOS Sleep Scale scores | Baseline and 4-6 weeks (estimated end of radiotherapy treatment)
  Change in MOS Sleep Scale scores between end of radiotherapy treatment and baseline

CONTACTS AND LOCATIONS:
Overall Officials: Ana Mañas, MD, Study Director — IMONCOLOGY, Hospital la Milagrosa. Madrid
Locations (11):
- Spain (11):
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela, A Coruña
  - Hospital de Terrassa, Terrassa, Barcelona
  - Hospital Puerta de Hierro, Majadahonda, Madrid
  - Hospital Do Meixoeiro, Vigo, Pontevedra
  - Centro Oncológico de galicia, A Coruña
  - Hospital de l'Esperança, Barcelona
  - ICO Hospitalet, Barcelona
  - Hospital Ramón y Cajal, Madrid
  - Hospital La Paz, Madrid
  - Hospital Regional de Málaga, Málaga
  - Hospital Virgen Macarena, Seville

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hernanz de Lucas R, Nunez Fernandez M, Gomez-Caamano A, Morera Lopez R, Fortes de la Torre I, de la Torre Tomas A, Munoz-Garzon V, Lopez Bermudo C, Manas Rueda A. Quality of life in patients with breakthrough cancer pain in radiation oncology departments in Spain: the CAVIDIOR study. Future Oncol. 2021 Mar;17(8):943-954. doi: 10.2217/fon-2020-1063. Epub 2020 Dec 8. PMID 33289432